CLINICAL TRIAL: NCT02338414
Title: An Observational Study to Evaluate the Efficacy of Romiplostim Administered at Every Other Week in Adult Patients With Chronic Immune Thrombocytopenia (ITP) Who Attained Platelet Counts ≥ 50 x 109/L After Weekly Doses of Romiplostim
Brief Title: An Observational Study to Evaluate the Efficacy of Biweekly Romiplostim in Adult Patients With ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jun Ho Jang, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPT-I001
Record Dates: First submitted 2015-01-06; First posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romiplostim (Other): Patients receiving romiplostim due to ITP
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Subcutaneous Romiplostim (weekly injection) -> if titrated with maintaining PLT count between 50-200 x 10^9/L -> Subcutaneous Romiplostim (biweekly injection)
  Other Names: Nplate

SUMMARY:
The aim of this study is to evaluate the efficacy of romiplostim administered at every other week in ITP patients who attained stable platelet counts ≥ 50 x 109/L for 4 consecutive weeks after weekly doses of romiplostim.

DETAILED DESCRIPTION:
Regarding the determination of appropriate dose, it is well known that romiplostim resulted in dose-dependent increases in platelet counts, but required dose for raising platelet count is variable between individuals according to each patient's ability to eliminate serum romiplostim. Because of this variability, after administration of initial 1mcg/kg of romiplostim, dose adjustment is recommended based on the platelet response to given dose of romiplostim. However, the optimal dose interval of romiplostim has rarely been studied. In pivotal studies, romiplostim was administered on a weekly schedule, and based on these studies, one dose at every week is being widely used. In one study in which ITP patients received weekly subcutaneous doses of romiplostim at a range from 3 to 15mcg/kg, half life of romiplostim was estimated from 1 to 34 days, suggesting that lengthening the interval between doses more than a week can be potentially possible in some patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has an ability to provide written informed consent prior to participating to the study
2. Subject is male or female ≥ 18 years of age
3. Subject has a diagnosis of immune thrombocytopenia (ITP) per the American Society of Hematology guidelines.
4. Subject received at least 1 prior therapy for ITP including corticosteroids, immunoglobulin, or splenectomy, but had an insufficient response to any of these treatment (PLT count should be < 30x109/L before romiplostim initiation.)
5. If subject had ever received TPO receptor agonist before, the patient can participate this study only after 8 weeks' wash out period

Exclusion Criteria:

1. Subject has a history of hematological malignancy, myeloproliferative disorder, myelodysplastic syndrome (MDS), or bone marrow stem cell disorder
2. Subject has participated in any study evaluating PEG-rHuMGDF, recombinant human thrombopoietin (rHuTPO), or related platelet product within 8 weeks
3. Subject has a known hypersensitivity to any recombinant E coli-derived product
4. Subject has received any therapeutic drug or device that is not approved by the local regulatory health agency for any indication within 4 weeks of Screening
5. Subject is of reproductive potential and is not using adequate contraceptive precautions, in the judgment of the investigator
6. Subject is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of biweekly romiplostim (platelet counts ≥ 30 x 10^9/L) | up to 24 weeks
  To evaluate the proportion of patients who had platelet counts ≥ 30 x 109/L during 4 or more weeks with biweekly romiplostim

CONTACTS AND LOCATIONS:
Overall Officials: Jong Wook Lee, M.D., Principal Investigator — Seoul St. Mary's Hospital, The Catholic University of Korea